CLINICAL TRIAL: NCT07094191
Title: Comparative Acute Effects of Caffeine-Free Chicory and Arabica Coffee on Inflammatory and Metabolic Responses to Exercise in Healthy Men: A Randomized Crossover Trial
Brief Title: The Effects of Acute Chicory Coffee Consumption on Exercise Performance and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatma Özsel Özcan (Other)
Responsible Party: Sponsor-Investigator, Fatma Özsel Özcan, Assistant Professor, Halic University
Organization: Halic University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2015-KAEK-79-23-03
Record Dates: First submitted 2025-07-21; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Fat Metabolism; Sport Nutrition; Exercise Metabolism; Inflammation; Glucose Metabolism
Keywords: arabica coffee; chicory coffee; metabolism; Inflammation; Plant-based ergogenic aids
MeSH Terms: conditions — Inflammation | interventions — METAL1 protein, Coffea arabica

STUDY DESIGN:
Intervention Model Description: This study used a single-blind, randomized, controlled, crossover design in which each participant received all three interventions (chicory coffee, arabica coffee, and control) in a randomized order. A 3-day washout period was implemented between each intervention to minimize carryover effects. The crossover model allowed within-subject comparisons of metabolic and performance responses to each beverage condition.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chicory Coffee Arm (Active Comparator): Participants in this arm consumed a standardized dose of chicory coffee (180 mL), a caffeine-free beverage rich in polyphenols and inulin, 45 minutes prior to the shuttle-run test. This arm was designed to assess the effects of chicory coffee on metabolism, inflammation, and exercise performance.
  Interventions: Dietary Supplement: Chicory Coffee (Caffeine-free, polyphenol-rich beverage from roasted chicory root)
- Arabica Coffee Arm (Active Comparator): Participants in this arm consumed a standardized dose of arabica coffee (180 mL), a regular caffeinated coffee, 45 minutes prior to the shuttle-run test. This arm served as a comparison to evaluate how caffeine-containing coffee influences metabolic and performance-related parameters.
  Interventions: Dietary Supplement: arabica coffee
- Control Arm (Other): CONTROL ARM
  Interventions: Dietary Supplement: no beverage control

INTERVENTIONS:
Dietary Supplement: Chicory Coffee (Caffeine-free, polyphenol-rich beverage from roasted chicory root) — A single oral dose of 180 mL chicory coffee prepared by steeping 20 grams of roasted and ground chicory root in hot water (approximately 90°C) for 5 minutes. The beverage was administered once, exactly 45 minutes before exercise, as part of a single session within a randomized crossover design. Chicory coffee is naturally caffeine-free, and rich in inulin and polyphenols, which are standardized in each preparation. No additional ingredients (milk, sugar, or flavoring) were added.
  Blood lactate, glucose, blood pressure, and oxygen saturation (SpO₂) levels were measured both before and after the exercise. In addition, venous blood samples were collected post-exercise to assess serum levels of adiponectin, interleukin-6 (IL-6), and tumor necrosis factor-alpha (TNF-α) and LPL.
  Arms: Chicory Coffee Arm
Dietary Supplement: arabica coffee — A single oral dose of 180 mL Arabica coffee prepared by steeping 20 grams of roasted and ground chicory root in hot water (approximately 90°C) for 5 minutes. The beverage was administered once, exactly 45 minutes before exercise, as part of a single session within a randomized crossover design. Chicory coffee is naturally caffeine-free, and rich in inulin and polyphenols, which are standardized in each preparation. No additional ingredients (milk, sugar, or flavoring) were added. Blood lactate, glucose, blood pressure, and oxygen saturation (SpO₂) levels were measured both before and after the exercise. In addition, venous blood samples were collected post-exercise to assess serum levels of adiponectin, interleukin-6 (IL-6), and tumor necrosis factor-alpha (TNF-α) and LPL.
  Arms: Arabica Coffee Arm
Dietary Supplement: no beverage control — Participants underwent the shuttle run exercise protocol in a fasted state, without consuming any food or beverages prior to the test. Blood lactate, glucose, blood pressure, and oxygen saturation (SpO₂) levels were measured both before and after the exercise. In addition, venous blood samples were collected post-exercise to assess serum levels of adiponectin, interleukin-6 (IL-6), and tumor necrosis factor-alpha (TNF-α) and LPL.
  Arms: Control Arm

SUMMARY:
The goal of this clinical trial is to evaluate the acute effects of chicory coffee on metabolism and exercise performance in healthy, moderately active male participants aged 18-25. The main questions it aims to answer are:

Does chicory coffee influence glucose, lipid, and energy metabolism after exercise?

Does chicory coffee affect physical performance and perceived fatigue levels?

Researchers will compare chicory coffee (CC), arabica coffee (AC), and a no-drink control to see if chicory coffee has similar or unique metabolic and performance effects compared to caffeinated coffee or no intervention.

Participants will:

Consume one of the test beverages (chicory coffee, arabica coffee, or no drink) 45 minutes before performing a shuttle-run test

Complete a standardized shuttle-run exercise test

Undergo blood sample collection before and after exercise to assess glucose, lactate, LPL, TNF-α, adiponectin, and IL-6

Rate their perceived exertion and record symptoms

DETAILED DESCRIPTION:
This study used a single-blind, randomized, controlled crossover design involving 22 healthy, moderately active male participants aged 18-25. Each participant underwent three intervention conditions in a randomized order:

Chicory coffee (CC)

Arabica coffee (AC)

Control (no beverage)

Before each trial, baseline data-including health status, dietary habits, and body composition-were collected. Participants consumed the assigned beverage 45 minutes before performing a shuttle-run test designed to assess endurance and physical performance. A 3-day washout period separated each intervention session to eliminate carryover effects.

During each session, pre- and post-exercise measurements included:

Blood glucose, lactate, blood pressure, and oxygen saturation

Subjective fatigue assessed by the Borg Rating of Perceived Exertion (RPE)

Additionally, venous blood samples were collected after exercise and analyzed for key metabolic and inflammatory biomarkers:

Lipoprotein lipase (LPL)

Tumor necrosis factor-alpha (TNF-α)

Adiponectin

Interleukin-6 (IL-6)

All blood samples were processed under cold-chain conditions and analyzed using ELISA methods. Dietary intake was monitored, and participants were instructed to maintain their usual eating habits while avoiding other caffeinated beverages during the study period.

Statistical analysis included MANOVA and ANOVA, with Bonferroni corrections used for multiple comparisons.

ELIGIBILITY:
Inclusion Criteria:

Male participants aged 18 to 25 years

Healthy status based on self-report and screening (no diagnosed chronic disease)

Moderately physically active (minimum 3 days/week of physical activity)

No regular use of medication or dietary supplements

Non-smoker

No caffeine consumption for at least 7 days prior to and during the study

Willing and able to provide informed consent

Able to complete the shuttle-run test as instructed

Exclusion Criteria:

Diagnosed with metabolic, cardiovascular, or inflammatory disease

Regular caffeine use or caffeine withdrawal symptoms

Use of alcohol, stimulants, or performance-enhancing substances during the study

Known allergy or intolerance to chicory or coffee

Participation in another clinical study within the last 30 days

Any musculoskeletal or respiratory condition that prevents safe participation in exercise

Inability to comply with the dietary or testing protocol

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05-18 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
This outcome measures blood lactate concentration in mmol/L to evaluate the metabolic response to shuttle run exercise. Capillary blood samples were taken from the fingertip at three time points: before, during, and immediately after exercise. | At baseline (immediately before exercise), mid-exercise, and immediately after exercise
  lactate measurement
Venous Blood Glucose Level | At baseline (pre-exercise) and within 10 minutes post-exercise
  This outcome measures venous blood glucose concentration (mg/dL) after completion of the shuttle run exercise protocol. Blood samples were collected from finger. Post-exercise glucose levels provide insight into glycemic regulation, insulin sensitivity, and metabolic response under fasting and exertional conditions.
Systolic and diastolic blood pressure | Systolic and diastolic blood pressure measured immediately before and immediately after exercise
  This outcome measures systolic and diastolic blood pressure (mmHg) to evaluate acute cardiovascular response to exercise. Measurements were taken at rest and immediately after the shuttle run using a digital sphygmomanometer.
Plasma Lipoprotein Lipase (LPL) Level (ng/mL) | At baseline and within 10 minutes post-exercise
  This outcome measures the concentration of plasma lipoprotein lipase (LPL) in ng/mL after completion of the shuttle run exercise protocol. Blood samples were collected post-exercise, and serum was analyzed to determine LPL levels using ELISA-based methods. This parameter reflects lipid metabolism activity in response to acute exercise under fasting conditions.
Subjective Fatigue Score (Borg Scale) | Immediately after completion of the shuttle run exercise protocol
  This outcome assesses perceived fatigue using the Borg Rating of Perceived Exertion (RPE) Scale immediately following the shuttle run exercise. Participants rated their level of physical exertion on a scale from 6 (no exertion at all) to 20 (maximal exertion). The Borg Scale is a validated tool for evaluating subjective fatigue and exercise intensity.
Tumor Necrosis Factor-alpha (TNF-α) | At baseline and within 10 minutes post-exercise
  This outcome measures the concentration of tumor necrosis factor-alpha (TNF-α) in serum samples collected after the shuttle run exercise protocol. TNF-α levels were analyzed using enzyme-linked immunosorbent assay (ELISA) techniques. TNF-α is a key pro-inflammatory cytokine, and its elevation post-exercise is indicative of acute inflammatory response and immune system activation.
Adiponectin | At baseline and within 10 minutes post-exercise
  This outcome measures the concentration of adiponectin in serum samples collected after the shuttle run exercise protocol. Serum adiponectin levels were determined using enzyme-linked immunosorbent assay (ELISA) methods. Adiponectin is an anti-inflammatory adipokine involved in glucose regulation and lipid metabolism, and its measurement provides insight into the metabolic response to acute exercise.
Interleukin-6 (IL-6) | At baseline and within 10 minutes post-exercise
  This outcome measures the concentration of interleukin-6 (IL-6) in serum samples collected after the shuttle run exercise protocol. IL-6 levels were determined using an enzyme-linked immunosorbent assay (ELISA). IL-6 is a pro-inflammatory cytokine known to respond acutely to physical exertion and is used as a biomarker of systemic inflammation and exercise-induced stress.

SECONDARY OUTCOMES:
Oxygen saturation | At baseline (immediately before exercise), mid-exercise, and immediately after exercise
  This outcome measures peripheral oxygen saturation (SpO₂) using a fingertip pulse oximeter. Measurements were taken at three time points: before, during, and immediately after the shuttle run exercise protocol. SpO₂ reflects the percentage of hemoglobin saturated with oxygen and is used to assess cardiopulmonary dynamics in response to physical exertion.

CONTACTS AND LOCATIONS:
Locations (1):
- Halic University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected in this study will not be made available to other researchers due to ethical considerations, limited scope of consent, and privacy protection of participants.

REFERENCES:
- [Background] Saunders TJ, Palombella A, McGuire KA, Janiszewski PM, Despres JP, Ross R. Acute exercise increases adiponectin levels in abdominally obese men. J Nutr Metab. 2012;2012:148729. doi: 10.1155/2012/148729. Epub 2012 May 30. PMID 22701167
- [Background] Yamashita K, Yatsuya H, Muramatsu T, Toyoshima H, Murohara T, Tamakoshi K. Association of coffee consumption with serum adiponectin, leptin, inflammation and metabolic markers in Japanese workers: a cross-sectional study. Nutr Diabetes. 2012 Apr 2;2(4):e33. doi: 10.1038/nutd.2012.6. PMID 23169586
- [Background] Diaz-Lara FJ, Del Coso J, Garcia JM, Portillo LJ, Areces F, Abian-Vicen J. Caffeine improves muscular performance in elite Brazilian Jiu-jitsu athletes. Eur J Sport Sci. 2016 Nov;16(8):1079-86. doi: 10.1080/17461391.2016.1143036. Epub 2016 Feb 10. PMID 26863885
- [Background] Bonnema AL, Kolberg LW, Thomas W, Slavin JL. Gastrointestinal tolerance of chicory inulin products. J Am Diet Assoc. 2010 Jun;110(6):865-8. doi: 10.1016/j.jada.2010.03.025. PMID 20497775